CLINICAL TRIAL: NCT05664399
Title: Shock Factor: Effects of Surprise on Cardiovascular Responses.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: HE2022-0286
Record Dates: First submitted 2022-12-05; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Physiologic Responses to Surprise Events
Keywords: Shock response; Ventilatory response; Cardiac response

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surprise events — Subjects will be subjected to 4 surprise events, two using Virtual Reality simulations of falling out of a boat, and 2 involving falling into dunk tanks of cool and thermoneutral water.

SUMMARY:
This research will determine the breathing, heart rate and other responses to four surprise events. For two events, virtual reality goggles will be used to create a realistic experience of falling out of a boat and rolling out of a boat or falling of a paddleboard. Two final events will involve falling into a dunk tank with either cool (20℃) or cold (10℃) water.

DETAILED DESCRIPTION:
Participants will participate in one visit to our research facility for 60-90 minutes. During this visit, the following will occur:

General overview

1. You will be considered for participation if you respond to the recruitment email from your organization, with an email to indicate interest in participation.
2. You will be sent an initial email asking if you would be willing to receive 4 files related to the study: They are Screening Questionnaire; Subject Information Form, Get Active Questionnaire; and Informed Consent.
3. If you respond positively to the second email you will be scheduled to appear at the research facility for an experimental trial.
4. Once you have arrived at the facility you will be asked to sign this Informed Consent Form if you have not already submitted it via email.
5. You will be asked if you voluntarily agree to be video recorded for the creation of educational videos for public use. If you do agree, you will be asked to sign a separate Audio-Video Release.
6. A pre-trial interview will be conducted, and responses will be manually recorded on paper.
7. You will then put on a special shirt (Hexoskin Shirt) over your swimsuit. This suit measures heart rate and breathing (indicated by the expansion of your chest).
8. You will then put on a climbing harness.
9. You will then complete 4 surprise events (see below in the Surprise Events section).
10. A post-trial interview will be conducted, and responses will be manually recorded.
11. You will change into your regular clothing and be free to leave the research facility.

Surprise Events

1. The first two events will involve wearing virtual reality (VR) goggles. The goggles will have visual presentations that coincide with the corresponding events that you are participating in. You will also wear a full climbing harness (including a chest harness) which is connected via climbing rope to a self-ratcheting lifeline that is firmly anchored to an overhead beam. The lifeline is commonly used to provide fall protection for workers at height; when the wearer falls, you will be slowly lowered to the ground. With this configuration, when you quickly rotate sideways or fall forward, you will experience the initial surprise motion, but your fall will be arrested by the lifeline. As an added safety measure, a gymnastics mat will be placed on the floor.

   1. For the first event, you will complete one of the following. you will either sit or stand on platforms that are initially stable but will then be allowed to rotate without notice (to simulate tipping a boat or falling off a standup paddleboard).
   2. For the second event, you will stand on the floor and either hold on to a rope (to simulate holding on to an anchor) or a fishing net (to simulate landing a fish). Without notice, either the rope or fishing net will be quickly pulled downwards.

   A movable gantry unit (overhead beam) will be used for these first two events. In each case, the self-ratcheting lifeline will be attached to the gantry, and the rope from the lifeline will be attached to the attachment on the back of the climbing harness; this will prevent you from ever falling to the ground.
2. The third and fourth events will not involve VR goggles but will involve falling into two dunk tanks with different water temperatures (cool = 22℃; cold = 10℃). The order of temperatures will be randomly assigned to achieve a balanced design. Before each dunking, you will shower in warm water so that your clothing is wet before both dunkings. You will then sit on the platform above one of the tanks. Once you are ready, without notice the dunk tank will be activated and you will be dunked and immediately allowed to exit. After about 5 minutes, the process will then be repeated for the second tank.

ELIGIBILITY:
Inclusion Criteria:

* Male and female boaters (anyone who takes 2 or more boat trips per year in small recreational boats (including powered and unpowered),
* 18-65 years old,
* healthy,
* do not have any allergic responses to water (aquagenic urticaria) or cold (cold urticaria),
* do not have a history of uncontrolled panic in water, or phobia or water (aquaphobia), and
* are cleared based on responses to the Get Active Questionnaire.
* Subjects will not have to be swimmers

Exclusion Criteria:

* Anyone who has a history of uncontrolled panic in water, or phobia of water (aquaphobia),
* allergic responses to water (aquagenic urticaria) or cold (cold urticaria),
* outside the 18-65 year old age bracket, and
* not cleared based on responses to the Get Active Questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female boaters (anyone who takes 2 or more boat trips per year in small recreational boats (including powered and unpowered), 18-65 years old and healthy.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory response | 1 day
  Changes in ventilation
Cardiac response | 1 day
  Changes in heart rate

SECONDARY OUTCOMES:
Subjective response | 1 day
  Subjective description of surprise experiences

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Giesbrecht, PhD, Principal Investigator — University of Manitoba
Locations (1):
- PlaySafe Productions, Keswick, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No